CLINICAL TRIAL: NCT03616756
Title: Fostering Resilience Amongst Mothers Under Stress: Authentic Connections for Nurse Leaders
Brief Title: Authentic Connections for Nurse Leaders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Sherry S. Chesak, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-002750
Record Dates: First submitted 2018-07-25; First posted 2018-08-06 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Stress
Keywords: Nurse leader; Resilience; Parenting; Stress; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Authentic Connections
- Control group (Active Comparator)
  Interventions: Behavioral: Protected time

INTERVENTIONS:
Behavioral: Authentic Connections — Authentic Connections support groups for nurse leaders who are also mothers. Meetings occur once a week for one hour.
  Arms: Intervention group
Behavioral: Protected time — Participants have one hour per week protected time scheduled on their calendar to do with what they choose.
  Arms: Control group

SUMMARY:
The purpose of this pilot study is to test the feasibility and outcomes of a supportive group-based intervention, Authentic Connections, to be used for nurse leaders at Mayo Clinic, Rochester, in a collaboration involving faculty at Arizona State University (ASU) Department of Psychology, Dr. Sunyia Luthar.

ELIGIBILITY:
* In an Nursing Education Specialist (NES) or Clinical Nurse Specialist (CNS) nurse leader role at Mayo Clinic Rochester
* Female gender
* A mother to at least one child or adult child

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Connor-Davidson Resilience Scale - 2 item | Baseline
  Two item scale, each of which has a 5-point range of responses, as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4). The total score ranges from 0-8, with higher scores reflecting greater resilience.
Connor-Davidson Resilience Scale - 2 item | 12 weeks
  Two item scale, each of which has a 5-point range of responses, as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4). The total score ranges from 0-8, with higher scores reflecting greater resilience.
Connor-Davidson Resilience Scale - 2 item | 24 weeks
  Two item scale, each of which has a 5-point range of responses, as follows: not true at all (0), rarely true (1), sometimes true (2), often true (3), and true nearly all of the time (4). The total score ranges from 0-8, with higher scores reflecting greater resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry S Chesak, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials